CLINICAL TRIAL: NCT04795232
Title: Recovery Kinetics Following Change of Direction (COD) Training in Soccer: Implications for Different COD Angles
Brief Title: Recovery Kinetics Following Change of Direction Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Recovery-COD Training-UTH
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Skeletal Muscle Damage
Keywords: change of direction training; recovery; soccer; performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in this arm will receive no intervention
- COD45 (Experimental): Participants in this arm will participate in a COD training session consisted of 45 degrees changes of direction
  Interventions: Other: COD45
- COD90 (Experimental): Participants in this arm will participate in a COD training session consisted of 90 degrees changes of direction
  Interventions: Other: COD90

INTERVENTIONS:
Other: COD45 — Participants will perform 2 sets of 10 sprints. The total distance for each sprint will be 27.6 meters and will include two changes of direction of 45 degrees. The recovery time will be 16 seconds between sprints and 2.20 minutes between sets
  Arms: COD45
Other: COD90 — Participants will perform 2 sets of 10 sprints. The total distance for each sprint will be 21.2 meters and will include two changes of direction of 90 degrees. The recovery time will be 16 seconds between sprints and 2.20 minutes between sets
  Arms: COD90

SUMMARY:
This study aims at investigating the recovery kinetics of skeletal muscle damage, neuromuscular fatigue and performance following a single change of direction (COD) training session in competitive soccer players. The impact of COD degrees will be also examined by comparing a 45o vs. 90o COD training session. Ten male soccer players will perform a COD45 [A single training session including 2x(10x ~27.6m) sprints with two 45o COD in each sprint], a COD90 [A single training session including 2x(10x ~21.2m) sprints with two 90o COD in each sprint] and a Control trial (No intervention included, only daily measurements) in randomized, repeated measures, crossover design. Assessments related to skeletal muscle damage, neuromuscular fatigue and performance will be performed prior to training session and daily for three consecutive days post-training, in each trial.

DETAILED DESCRIPTION:
Ten male soccer players will be included in this study. Participants will be initially informed about the aim of study as well as the associated risks and benefits and subsequently will provide their signed consent form. At baseline, they will undergo assessment of their anthropometrics (i.e. body mass and body height), body composition (by DXA), physical conditioning status [maximal oxygen consumption (VO2max), Yo-Yo Intermittent Endurance test level 2 and Yo-Yo Intermittent Recovery test level 2] and daily dietary intake. Thereafter, they will participate in two experimental trials and one control trial in a randomized, crossover, repeated measures design: i) COD45: Participants in this trial will perform a COD training session consisted of 2 sets of 10 x ~27.6m sprints with two 45o COD in each sprint and a resting period of 16 sec and 2:20 min between sprints and sets, respectively, ii) COD90: Participants in this trial will perform a COD training session consisted of 2 sets of 10 x ~21.2m sprints with two 90o COD in each sprint and a resting period of 16 sec and 2:20 min between sprints and sets, respectively, iii) Control: Participants in this trial will only participate in daily assessments to control for day to day variability in the depended variables (they will not receive any intervention). Prior to each trial, participants will provide a resting blood sample (for the determination of blood lactate, white blood cell count and creatine kinase activity) and undergo assessment of their delayed onset of muscle soreness (DOMS), maximal voluntary isometric contraction (MVIC), countermovement jump [will be assessed using two force platforms at 1000 Hz and electromyography instrumentation (EMG)], isokinetic peak torque of knee extensors and flexors (will be assessed on an isokinetic dynamometer), agility (will be assessed using the Illinois test), 10m and 30m sprint time (will be assessed by using light cells) and repeated sprint ability (5x30m sprints will be performed with 25 sec rest in-between). In COD45 and COD90 experimental trials, a blood sample will be collected immediately post-training for the determination of blood lactate concentration while assessment of DOMS, MVIC and countermovement jump will be performed at 1, 2 and 3 hours post-training. In all trials assessment of DOMS, MVIC, countermovement jump (CMJ), isokinetic peak torque, agility and sprinting performance as well as determination of creatine kinase activity and white blood cell count will be performed at 24, 48 and 72 hours post-training. A 7-day wash out period will applied between trials.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players participating in at least 5 training sessions per week and 1official match
* Participation at a competitive level for at least 4 years
* Free of musculoskeletal injuries
* No use of ergogenic supplements or medication
* Non-smokers

Exclusion Criteria:

* Musculoskeletal injury
* Use of alcohol, caffeine and any type of ergogenic supplements or medication during the course of the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in creatine kinase activity | At baseline, at 24, 48 and 72 hours after change of direction training session
  Creatine kinase activity will be measured in plasma
Change in white blood cell count | At baseline, at 24, 48 and 72 hours after change of direction training session
  White blood cell count will be measured by using an automatic blood analyzer
Change in delayed onset of muscle soreness | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Muscle soreness will be assessed by palpation of the muscle belly and the distal region
Change in isometric peak torque | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Isometric peak torque will be assessed on an isokinetic dynamometer
Change in fatigue index of maximal voluntary isometric contraction during 10 seconds | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Fatigue rate will be determined by calculating the percent drop of peak torque between the first and the last three seconds of a 10-second maximal isometric contraction
Change in isokinetic peak torque of knee extensors | At baseline, at 24, 48 and 72 hours after change of direction training session
  Isokinetic peak torque will be assessed on an isokinetic dynamometer in both limbs
Change in isokinetic peak torque of knee flexors | At baseline, at 24, 48 and 72 hours after change of direction training session
  Isokinetic peak torque will be assessed on an isokinetic dynamometer in both limbs
Change in countermovement jump height | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Countermovement jump height will be assessed by using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height for each leg
Change in ground reaction force during countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Ground reaction force will be assessed by using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height for each leg
Change in peak power during countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Peak power will be assessed using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height for each leg
Change in mean power during countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Mean power will be assessed using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height for each leg
Change in vertical stiffness during countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Vertical stiffness will be assessed using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height for each leg
Change in peak rate of force development during countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  Peak rate of force development will be assessed using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height for each leg
Change in peak normalized electromyography (EMG) during the eccentric and concentric phases of the countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  EMG data will be collected wirelessly at 2000 Hz using a Myon MA-320 EMG system (Myon AG, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius and gluteus maximus muscles.
Change in mean normalized electromyography (EMG) during the eccentric and concentric phases of the countermovement jump | At baseline, at 1, 2, 3, 24, 48 and 72 hours after change of direction training session
  EMG data will be collected wirelessly at 2000 Hz using a Myon MA-320 EMG system (Myon AG, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius and gluteus maximus muscles.
Change in repeated sprint ability | At baseline, at 24, 48 and 72 hours after change of direction training session
  Repeated sprint ability will be tested using 5x30 m sprints with 25 seconds rest in-between
Change in sprint time of 10m | At baseline, at 24, 48 and 72 hours after change of direction training session
  10m sprint time will be assessed using light cells
Change in sprint time of 30m | At baseline, at 24, 48 and 72 hours after change of direction training session
  30m sprint time will be assessed using light cells
Change in agility | At baseline, at 24, 48 and 72 hours after change of direction training session
  Agility will be assessed using the illinois agility test.
Change in field activity during the change of direction training session | During the change of direction training session
  Field activity will be continuously monitored during the change of direction training session by using global positioning system (GPS)
Change in heart rate during the change of direction training session | During the change of direction training session
  Heart rate will be continuously monitored during the change of direction training session by using heart rate monitors.
Change in blood lactate concentration | At baseline and immediately post change of direction training session
  Blood lactate will be measured using a lactate plus system

SECONDARY OUTCOMES:
Body mass | At baseline
  Body mass will me measured on a beam balance with stadiometer
Body height | At baseline
  Body height will me measured on a beam balance with stadiometer
Body fat | At baseline
  Body fat will be assessed by using Dual-emission X-ray absorptiometry
Lean body mass | At baseline
  Lean body mass will be assessed by using Dual-emission X-ray absorptiometry
Maximal oxygen consumption (VO2max) | At baseline
  VO2max will be measured by open circuit spirometry via breath by breath method
Yo-Yo Intermittent Endurance Test level 2 performance | At baseline
Yo-Yo Intermittent Recovery Test level 2 performance | At baseline
Dietary intake | At baseline
  Dietary intake will be assessed over a 7-day period by using diet recalls

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Prof, Study Director — University of Thessaly, Department of Physical Education and Sport Science
Locations (2):
- Greece (2):
  - SMART LAB, Department of Physical Education and Sports Science, University of Thessaly., Trikala
  - SmArT LABORATORY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES, UNIVERSITY OF THESSALY, Trikala

IPD SHARING:
Plan to Share IPD: No